CLINICAL TRIAL: NCT00537381
Title: A Randomized, Double-blind, Multicenter, Phase 2 Study of a Human Monoclonal Antibody to Human av Integrins (CNTO 95) in Combination With Docetaxel for the First-Line Treatment of Subjects With Metastatic Hormone Refractory Prostate Cancer
Brief Title: An Efficacy and Safety Study of Intetumumab (CNTO 95) in Participants With Metastatic Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013249; C1034T08 (Other: Centocor, Inc.); 2006-005766-39 (EudraCT Number)
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; CNTO 95; Intetumumab; Docetaxel; Prednisone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; intetumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel + Prednisone + Placebo (Active Comparator): Matching placebo as intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) every week for initial 6 weeks, then every 3 weeks; along with docetaxel 75 milligram per square meter (mg/m^2) as intravenous infusion every 3 weeks and prednisone 5 mg orally twice daily were administered till 6 months or disease progression.
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Placebo
- Docetaxel + Prednisone + Intetumumab (Experimental): Intetumumab 10 mg per kilogram (mg/kg) as intravenous infusion every week for initial 6 weeks, then every 3 weeks; along with docetaxel 75 mg/m^2 as intravenous infusion every 3 weeks and prednisone 5 mg orally twice daily were administered till 6 months or disease progression.
  Interventions: Drug: Docetaxel; Drug: Prednisone; Biological: Intetumumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m^2 as intravenous infusion every 3 weeks.
Drug: Prednisone — Prednisone 5 mg orally twice daily.
Biological: Intetumumab — Intetumumab 10 mg/kg as intravenous infusion every week for initial 6 weeks, then every 3 weeks.
  Other Names: CNTO 95
  Arms: Docetaxel + Prednisone + Intetumumab
Drug: Placebo — Placebo matching to intetumumab, as intravenous infusion every week for initial 6 weeks, then every 3 weeks.
  Arms: Docetaxel + Prednisone + Placebo

SUMMARY:
The purpose of this study is to assess the effects of intetumumab when given in combination with docetaxel and prednisone to participants with metastatic (spread of cancer cells from one part of the body to another) hormone-refractory (not responding to treatment) prostate cancer (abnormal tissue that grows and spreads in the body until it kills).

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), randomized (the study drug is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives) study of intetumumab in combination with docetaxel and prednisone for the first-line treatment of participants with metastatic hormone-refractory prostate cancer. There will be 2 study groups. One group will receive intetumumab in combination with docetaxel and prednisone (study treatment) and the other group will receive placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) matching to intetumumab in combination with docetaxel and prednisone (control treatment). The duration of treatment will be 6 months. Participants who respond to treatment with stable disease or better will receive extended treatment until disease progression (disease worsening) or for an additional 6 months, whichever occurs first. Treatment can be further continued with the sponsor's discretion after receiving 6 months of extended treatment, if participant response to the treatment (with stable disease, partial response, or complete response). Participants who have confirmed progressive disease while receiving study treatment may have their treatment unblinded (participants will know the name of drug which was given to them), if they wish to be considered for alternative treatment. Participants who were receiving the control treatment will be considered to have completed the study treatment, and will have the option to receive alternative treatment. Alternative treatment will either be intetumumab along with docetaxel and prednisone or intetumumab alone. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria

* Confirmed cancer of the prostate
* Evidence of metastatic disease
* Have a life expectancy greater than 12 weeks
* Have at least 4 weeks from previous major surgery to date of first study agent given
* Have progressive hormone-refractory disease after orchiectomy or gonadotropin-releasing hormone analog and/or antiandrogen treatment within 6 months prior to the first study agent administration Exclusion Criteria
* Have known Central Nervous System metastases (cancerous tumors that have spread to the brain from somewhere else in the body)
* Had prior systemic non-hormonal therapy for hormone refractory prostate cancer
* Have known Human Immunodeficiency Virus (HIV, a life-threatening infection which you can get from an infected person's blood or from having sex with an infected person) seropositivity or known hepatitis B or C infection
* Have planned major surgery during the study
* Have taken any over-the-counter (medicine that can be bought without a prescription) or herbal treatment for prostate cancer within 4 weeks prior to the first study treatment administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (59):
- United States (7):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Bernardino, California
  - Wichita, Kansas
  - Shreveport, Louisiana
  - Charleston, South Carolina
  - North Charleston, South Carolina
- Austria (3):
  - Graz
  - Vienna
  - Wels
- Belgium (10):
  - Antwerp
  - Brasschaat
  - Brussels
  - Haine-Saint-Paul, La Louviere
  - Leuven
  - Liÿge
  - Ottignies
  - Roeselare
  - Tournai
  - Wilrijk
- Germany (8):
  - Aschaffenburg
  - Berlin
  - Cologne
  - Freiburg im Breisgau
  - Kirchheim
  - Marburg
  - München
  - Tübingen
- India (6):
  - Ahmedabad
  - Bangalore
  - Chennai
  - Mumbai
  - New Delhi
  - Pune
- Netherlands (5):
  - Apeldoorn
  - Leiden
  - Maastricht
  - Nijmegen
  - The Hague
- Poland (6):
  - Bydgoszcz
  - Gdansk
  - Inowrocław
  - Kościerzyna
  - Lodz
  - Lublin
- Russia (7):
  - Moscow
  - Moscow Region
  - Saint Petersburg
  - St-Petersburg Leningrad
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- South Africa (3):
  - Johannesburg Gauteng
  - Pretoria
  - Pretoria Gauteng
- United Kingdom (4):
  - Cambridge
  - Leicester
  - Lincoln
  - London

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel + Prednisone + Placebo: Matching placebo as intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) every week for initial 6 weeks, then every 3 weeks; along with docetaxel 75 milligram per square meter (mg/m^2) as intravenous infusion every 3 weeks and prednisone 5 mg orally twice daily were administered till 6 months or disease progression. Participants with disease progression at any time had option to crossover to alternative treatment with intetumumab alone or intetumumab in combination with docetaxel and prednisone.
Period: Overall Study
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Started | 65 (11 Participants after disease progression switched to intetumumab alone (2) or D+P+ Intetumumab (9).) | 66
Completed | 9 | 4
Not Completed | 56 | 62
Not completed — Adverse Event | 13 | 9
Not completed — Death | 3 | 3
Not completed — Withdrawal by Subject | 5 | 14
Not completed — Physician Decision | 7 | 6
Not completed — Disease Progression | 9 | 18
Not completed — Sponsor decision | 14 | 9
Not completed — Other | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel + Prednisone + Placebo: Matching placebo as intravenous infusion every week for initial 6 weeks, then every 3 weeks; along with docetaxel 75 milligram per square meter (mg/m^2) as intravenous infusion every 3 weeks and prednisone 5 mg orally twice daily were administered till 6 months or disease progression. Participants with disease progression at any time had option to crossover to alternative treatment with intetumumab alone or intetumumab in combination with docetaxel and prednisone.
- Total: Total of all reporting groups
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab | Total
Number analyzed (Participants) | 65 | 66 | 131
Age Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (8.74) | 66.3 (7.51) | 66.7 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 65 | 66 | 131
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 3 | 2 | 5
  BELGIUM | 10 | 9 | 19
  GERMANY | 19 | 14 | 33
  INDIA | 11 | 10 | 21
  NETHERLANDS | 2 | 5 | 7
  POLAND | 13 | 10 | 23
  RUSSIAN FEDERATION | 4 | 12 | 16
  SOUTH AFRICA | 1 | 0 | 1
  UNITED KINGDOM | 1 | 1 | 2
  UNITED STATES | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The PFS was assessed as median number of days from baseline until the first documented sign of disease progression (increase in disease; radiographic, clinical, or both) or death due to any cause, whichever occurred earlier.
Time Frame: Baseline up to 6 months after last dose of study treatment, assessed up to 551 days
Population: Efficacy population included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Number analyzed (Participants) | 65 | 66
Days | 336.0 [266.0 to 477.0] | 232.0 [155.0 to 320.0]
Statistical Analysis 1: Comparison: Docetaxel + Prednisone + Placebo vs Docetaxel + Prednisone + Intetumumab; Test type: Superiority or Other; p = 0.014, Log Rank; Hazard Ratio (HR) = 1.728, 95% CI 2-sided [1.112 to 2.686] — Hazard ratio and 95% confidence interval was estimated from a Cox proportional hazards model with treatment as the only explanatory factor

2. Secondary Outcome: Number of Participants With Best Overall Response (OR)
Description: Number of participants with best OR is based on assessment of confirmed complete response (CR) or confirmed partial response (PR). Confirmed CR is defined as disappearance of all target lesions. Confirmed PR is defined as greater than or equal to 30 percent decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD. Confirmed responses are those that persist on repeat imaging study greater than or equal to 4 weeks after initial documentation of response.
Time Frame: Baseline up to 6 months after last dose of study treatment, assessed up to 551 days
Population: Response evaluable population included participants who had target lesion or non-target lesion at baseline and received at least 1 study treatment and had at least 1 post-baseline response assessment or discontinued study treatment due to disease progression, or death.
Measure: Number; unit: Participants
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Number analyzed (Participants) | 50 | 50
Participants
  Complete Response | 1 | 0
  Partial Response | 9 | 8
Statistical Analysis 1: Comparison: Docetaxel + Prednisone + Placebo vs Docetaxel + Prednisone + Intetumumab; Test type: Superiority or Other; p = 0.795, Fisher Exact

3. Secondary Outcome: Number of Participants With Prostate Specific Antigen (PSA) Response
Description: The PSA response is defined as at least a 50 percent decrease in PSA below the baseline value, confirmed by a second PSA value greater than or equal to 6 weeks later. A participant was considered to be a PSA responder if and only if the response occurs prior to PSA progression (increase of at least 25 percent and an increase of 5 nanogram per milliliter from the lowest observed PSA value since initiation of treatment, to be confirmed greater than or equal to 3 weeks later).
Time Frame: Baseline up to 6 months after last dose of study treatment or early withdrawal, assessed up to 601 days
Population: Included all participants randomly assigned to study treatment and had baseline PSA evaluation and at least two post-baseline evaluations that are at least 3 weeks apart.
Measure: Number; unit: Participants
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Number analyzed (Participants) | 63 | 58
Participants | 43 | 27
Statistical Analysis 1: Comparison: Docetaxel + Prednisone + Placebo vs Docetaxel + Prednisone + Intetumumab; Test type: Superiority or Other; p = 0.018, Fisher Exact

4. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from the date of randomization to death due to any cause. For participants who were alive at the time of analysis, overall survival was censored at the last contact date.
Time Frame: Baseline until death (up to 887 days)
Population: Efficacy population included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Number analyzed (Participants) | 65 | 66
Days | 626.0 [532.0 to NA] — Upper limit of confidence interval was not estimable due to the high number of participants censored for survival. | 522.0 [418.0 to NA] — Upper limit of confidence interval was not estimable due to the high number of participants censored for survival.
Statistical Analysis 1: Comparison: Docetaxel + Prednisone + Placebo vs Docetaxel + Prednisone + Intetumumab; Test type: Superiority or Other; p = 0.163, Log Rank; Hazard Ratio (HR) = 1.476, 95% CI 2-sided [0.853 to 2.522] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percent Change From Baseline in 'C-telopeptide of Type I Collagen (CTx)' Marker Concentration
Description: Percent change = marker concentration at time of measurement minus baseline value divided by baseline value multiplied by 100.
Time Frame: Baseline, Week 6, 7, 10 and 13
Population: The pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study treatment and had at least 1 PD measurement. Here 'n' signifies those participants evaluable for this measure at the specified time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Number analyzed (Participants) | 11 | 65
Percent change
  Percent Change at Week 6 (n = 10, 48) | 1.45 (51.019) | -30.81 (42.091)
  Percent Change at Week 7 (n = 10, 54) | -11.58 (45.396) | -39.78 (32.437)
  Percent Change at Week 10 (n = 11, 51) | 2.39 (53.537) | -25.48 (122.178)
  Percent Change at Week 13 (n = 11, 41) | 5.22 (59.728) | -44.89 (40.941)

6. Secondary Outcome: Percent Change From Baseline in 'N-telopeptide of Type I Collagen (NTx)' Marker Concentration
Description: as for outcome 5
Time Frame: Baseline, Week 6, 7, 10 and 13
Population: The PD analysis set included all participants who received at least 1 dose of study treatment and had at least 1 PD measurement. Here 'n' signifies those participants evaluable for this measure at the specified time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Number analyzed (Participants) | 11 | 65
Percent change
  Percent Change at Week 6 (n = 10, 48) | -0.77 (37.584) | -21.37 (47.747)
  Percent Change at Week 7 (n = 10, 54) | 1.58 (40.651) | -23.44 (34.703)
  Percent Change at Week 10 (n = 11, 51) | 2.55 (46.433) | -21.71 (63.890)
  Percent Change at Week 13 (n = 11, 40) | -3.87 (31.845) | -36.47 (25.701)

7. Secondary Outcome: Percent Change From Baseline in 'Vascular Endothelial Growth Factor (VEGF)' Marker Concentration
Description: as for outcome 5
Time Frame: Baseline, Week 6, 7, 10 and 13
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab
Number analyzed (Participants) | 11 | 65
Percent change
  Percent Change at Week 6 (n = 10, 48) | -10.00 (29.609) | -9.64 (34.229)
  Percent Change at Week 7 (n = 10, 54) | -3.10 (24.465) | 11.69 (41.338)
  Percent Change at Week 10 (n = 11, 51) | 3.96 (27.859) | 32.11 (85.953)
  Percent Change at Week 13 (n = 11, 41) | 8.22 (32.622) | 20.19 (55.565)

ADVERSE EVENTS:
Groups:
- Docetaxel + Prednisone + Placebo/ Intetumumab: Participants who initially received Docetaxel + Prednisone + Placebo until disease progression were switched their treatment to intetumumab alone (2 participants) and received intetumumab 10 mg/kg as intravenous infusion every 3 weeks till disease progression.
- Docetaxel + Prednisone + Placebo/ D+ P + Intetumumab: Participants who initially received Docetaxel + Prednisone + Placebo until disease progression were switched their treatment to Docetaxel (D) + Prednisone (P) + intetumumab (9 participants) and received intetumumab 10 mg/kg as intravenous infusion every 3 weeks; along with docetaxel 75 mg/m^2 as intravenous infusion every 3 weeks and prednisone 5 mg orally twice daily till disease progression.
Arm/Group | Docetaxel + Prednisone + Placebo | Docetaxel + Prednisone + Intetumumab | Docetaxel + Prednisone + Placebo/ Intetumumab | Docetaxel + Prednisone + Placebo/ D+ P + Intetumumab
Serious Adverse Events (participants affected / at risk) | 23/65 | 24/66 | 1/2 | 4/9
Other Adverse Events (participants affected / at risk) | 59/65 | 59/66 | 2/2 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Prednisone + Placebo (N=65) | Docetaxel + Prednisone + Intetumumab (N=66) | Docetaxel + Prednisone + Placebo/ Intetumumab (N=2) | Docetaxel + Prednisone + Placebo/ D+ P + Intetumumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 2 | 3 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1
Extravasation (General disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Coagulation time prolonged (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 3 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Pneumatic compression therapy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Prednisone + Placebo (N=65) | Docetaxel + Prednisone + Intetumumab (N=66) | Docetaxel + Prednisone + Placebo/ Intetumumab (N=2) | Docetaxel + Prednisone + Placebo/ D+ P + Intetumumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 12 | 9 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 22 | 16 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 21 | 14 | 0 | 1
Dry eye (Eye disorders) | 4 | 3 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 5 | 2 | 0 | 0
Lacrimation increased (Eye disorders) | 8 | 7 | 0 | 2
Ocular hyperaemia (Eye disorders) | 1 | 4 | 0 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 4 | 0 | 0
Vision blurred (Eye disorders) | 4 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 13 | 9 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 22 | 18 | 0 | 2
Gastritis (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 17 | 18 | 1 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 9 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 10 | 6 | 1 | 0
Asthenia (General disorders) | 16 | 15 | 1 | 0
Fatigue (General disorders) | 17 | 17 | 0 | 2
Hypothermia (General disorders) | 4 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 4 | 2 | 0 | 0
Oedema peripheral (General disorders) | 7 | 8 | 0 | 0
Pain (General disorders) | 5 | 1 | 0 | 0
Pyrexia (General disorders) | 10 | 13 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 6 | 3 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Moraxella infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 2 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 9 | 1 | 1
Enzyme abnormality (Metabolism and nutrition disorders) | 4 | 5 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 9 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 4 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 3 | 0 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 7 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 7 | 6 | 0 | 0
Dysgeusia (Nervous system disorders) | 15 | 13 | 0 | 1
Headache (Nervous system disorders) | 9 | 13 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 10 | 11 | 0 | 1
Paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 9 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 7 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 8 | 1 | 2
Proteinuria (Renal and urinary disorders) | 4 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 17 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 9 | 7 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 12 | 7 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 0 | 0
Hypertension (Vascular disorders) | 5 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Treatment with intetumumab/placebo was permanently discontinued after a planned, preliminary review of interim analysis data. Therefore, study treatment with intetumumab was not completed for some participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less